CLINICAL TRIAL: NCT04733495
Title: A Group-Mediated Cognitive Behavioral Resistance Exercise Intervention in Head and Neck Cancer Patients Undergoing Chemoradiation Treatment
Brief Title: Group-Mediated Cognitive Behavioral Resistance Exercise Intervention in Head and Neck Cancer Patients Undergoing Chemoradiation Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Dukagjin Blakaj, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-19113; NCI-2020-13834 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-01-06; First posted 2021-02-02 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Locally Advanced Head and Neck Squamous Cell Carcinoma
MeSH Terms: interventions — Counseling; Nutrition Assessment; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (resistance exercise, counseling) (Experimental): Patients undergo personalized resistance exercises over 1 hour daily. Patients receive dietary counseling over 60 minutes at week 1 and then over 15-30 minutes weekly for up to 6 weeks. Patients also receive group-based behavioral counseling BIW in weeks 1-8, QW in weeks 9-12, and then twice a month in weeks 13-24.
  Interventions: Other: Counseling; Behavioral: Dietary Counseling and Surveillance; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Resistance Training

INTERVENTIONS:
Other: Counseling — Receive group-based behavioral counseling
  Other Names: Counseling Intervention
Behavioral: Dietary Counseling and Surveillance — Receive dietary counseling
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Other: Resistance Training — Undergo personalized resistance exercises
  Other Names: Strength Training

SUMMARY:
This clinical trial examines a group-mediated cognitive behavioral resistance exercise intervention in head and neck cancer patients who are undergoing chemoradiation treatment. Chemoradiation is the established standard of care for locally advanced head and neck cancer patients. However, many head and neck cancer patients experience clinically meaningful declines in muscle mass, physical function, and quality of life during and following treatment. Resistance exercise has been shown to improve muscle mass, body composition, and physical function when integrated with appropriate standard of care nutritional counseling/supplementation. This trial may help researchers determine the important of integrating exercise interventions with routine cancer care.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of implementing a group-mediated cognitive behavioral (GMCB) personalized resistance exercise (RE) intervention in head and neck cancer (HNCa) patients undergoing chemoradiation (CRT).

II. To examine the effects of GMCB RE intervention upon functional limitations, body composition, and quality of life (QOL) in HNCa patients undergoing CRT.

OUTLINE:

Patients undergo personalized resistance exercises over 1 hour daily. Patients receive dietary counseling over 60 minutes at week 1 and then over 15-30 minutes weekly for up to 6 weeks. Patients also receive group-based behavioral counseling twice weekly (BIW) in weeks 1-8, once a week (QW) in weeks 9-12, and then twice a month in weeks 13-24.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced human papillomavirus (HPV)+ stage III-IV head and neck (HN) squamous cell carcinomas undergoing concurrent chemotherapy and radiation therapy. Patients with prior cancers or post-surgical patients needing adjuvant therapy will not be allowed to participate in this study
* Undergoing planned course of standard of care CRT for a total of 33 to 35 RT fractions (six and a half or seven weeks of treatment)
* Adults 18 years old (yo) or older who have clearance from their primary care provider (PCP) or medical oncologist to participate in resistance exercises during treatment. These patients will be monitored very closely on a weekly basis during the trial
* All participants must be free of severe heart or systemic disease or medical contraindications that would make supervised RE participation unsafe
* Receive medical clearance to participate from treating primary care physician or Medical Oncologists
* Ability to understand and the willingness to sign a written informed consent
* Willing and physically able to participate in RE

Exclusion Criteria:

* Severe heart or systemic disease or medical contraindications to exercise
* Diagnosis of cancer other than HNCa
* Musculoskeletal/Neurological disorder inhibiting them from safe exercise
* Pregnant or nursing women
* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2022-05-22 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Recruitment rates | At baseline
  Number of patients agreed to participate by signing the informed consent
Adherence of Intervention | At 3-month
  Adherence will be defined via session attendance and compliance with the prescribed sets, repetitions, and loads of the RE prescription as assessed using exercise logs, upon which participants will record all exercise performed at the center or independently..
Adherence of Intervention | At 6-month
  Adherence will be defined via session attendance and compliance with the prescribed sets, repetitions, and loads of the RE prescription as assessed using exercise logs, upon which participants will record all exercise performed at the center or independently..
Incidence of adverse events | At 3-month
  Monitored by direct observation and or patient reporting of signs and symptoms using NCI CTCAE version 5
Incidence of adverse events | At 6-month
  Monitored by direct observation and or patient reporting of signs and symptoms using NCI CTCAE version 5
Retention rates | At 3-month
  Rates will be calculated prospectively throughout the trial
Retention rates | At 6-month
  Rates will be calculated prospectively throughout the trial
Functional Battery | At 3-month
  Functional Battery Objective Functional Performance will be assessed using 3 valid and reliable timed performance-related mobility tasks: 400-meter walk (the primary outcome), stair-climb, and lift and carry task. Assessments of Mobility-Related Self-Efficacy to complete each functional task will also be completed with the tests.
Functional Battery | At 6-month
  Functional Battery Objective Functional Performance will be assessed using 3 valid and reliable timed performance-related mobility tasks: 400-meter walk (the primary outcome), stair-climb, and lift and carry task. Assessments of Mobility-Related Self-Efficacy to complete each functional task will also be completed with the tests.
Patient Reported Outcomes (Quality of Life/Fatigue/Physical Function) | At 3-month
  QoF will be assessed using both global and disease-specific measures including the satisfaction with life scale, the SF-12, the Functional Assessment of Cancer Therapy - Head and Neck (FACT - HN) and the EORTC Quality of Life scale. Fatigue symptoms will be assessed with the Brief Fatigue Inventory (BFI).
Patient Reported Outcomes (Quality of Life/Fatigue/Physical Function) | At 6-month
  QoF will be assessed using both global and disease-specific measures including the satisfaction with life scale, the SF-12, the Functional Assessment of Cancer Therapy - Head and Neck (FACT - HN) and the EORTC Quality of Life scale. Fatigue symptoms will be assessed with the Brief Fatigue Inventory (BFI).
Muscular strength | At 3-month
  Muscular strength will be assessed using standardized one-repetition maximum testing protocols for the chest press and leg extension exercises.
Muscular strength | At 6-month
  Muscular strength will be assessed using standardized one-repetition maximum testing protocols for the chest press and leg extension exercises.
Anthropometric measurements | At 3-month
  Anthropometric measurements are a series of quantitative measurements of the muscle, bone, and adipose tissue used to assess the composition of the body. The core elements of anthropometry are height, weight, body mass index (BMI), body circumferences (waist, hip, and limbs), and skinfold thickness. Anthropometric measurements will be taken in a consultation room to ensure the privacy of the participant.
Anthropometric measurements | At 6-month
  Anthropometric measurements are a series of quantitative measurements of the muscle, bone, and adipose tissue used to assess the composition of the body. The core elements of anthropometry are height, weight, body mass index (BMI), body circumferences (waist, hip, and limbs), and skinfold thickness. Anthropometric measurements will be taken in a consultation room to ensure the privacy of the participant.
Body composition | At 3-month
  Body composition will be assessed using dual-energy x-ray absorptiometry (DEXA; GE Health Care Lunar, Madison, WI) for all outcome measures. The DEXA scans will be used to determine total body composition including bone-mineral density, as well as, percentage body fat and fat-free mass for all body regions.
Body composition | At 6-month
  Body composition will be assessed using dual-energy x-ray absorptiometry (DEXA; GE Health Care Lunar, Madison, WI) for all outcome measures. The DEXA scans will be used to determine total body composition including bone-mineral density, as well as, percentage body fat and fat-free mass for all body regions.

CONTACTS AND LOCATIONS:
Overall Officials: Dukagjin Blakaj, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

DOCUMENTS (1):
  • Informed Consent Form (2022-11-19): https://cdn.clinicaltrials.gov/large-docs/95/NCT04733495/ICF_000.pdf